CLINICAL TRIAL: NCT06844240
Title: Efficacy and Safety of the XEN63: a Prospective Observational Multicenter Study.
Brief Title: Efficacy and Safety of XEN63 Gel Implant
Acronym: XEN63
Status: Enrolling by invitation | Type: Observational
Sponsor: Mario Stirpe (Other)
Responsible Party: Sponsor-Investigator, Mario Stirpe, Prof, Fondazione G.B. Bietti, IRCCS
Organization: Fondazione G.B. Bietti, IRCCS (Other)
Other Study IDs: GLC06-23
Record Dates: First submitted 2025-01-31; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-01

CONDITIONS: Glaucoma
Keywords: glaucoma; surgery; XEN63
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Glaucoma: Diagnosis of primary or secondary open-angle glaucoma according to the diagnostic criteria of 4th edition of the European Glaucoma Society Guidelines.

SUMMARY:
The study is prospective, observational, multicenter and has the aim of evaluating the efficacy and safety of the XEN63 implant in patients with primary or secondary glaucoma who require surgery in association or not with cataract surgery, for IOP not controlled by medical therapy, disease progression or intolerance to topical therapy, comparing IOP values before and 24 months after implantation.

DETAILED DESCRIPTION:
The study is prospective, observational, multicenter and has the aim of evaluating the efficacy and safety of the XEN63 implant in patients with primary or secondary glaucoma who require surgery in association or not with cataract surgery, for IOP not controlled by medical therapy, disease progression or intolerance to topical therapy, comparing IOP values before and 24 months after implantation. Every patients will be followed for 24 months.

Secondary aims of the study are:

* Evaluating the hypotensive efficacy of the XEN63 12 months after implantation.
* Assessing the safety of the XEN63 device after 12 and 24 months after implantation.
* Comparing the hypotensive efficacy of the XEN63 in glaucomatous patients undergoing the solo procedure and in those undergoing the combo procedure
* Evaluating the quality of life of patients undergoing XEN63 implantation 12 and 24 months after implantation.
* Evaluating the association between factors related to the patient, the surgical technique or post-operative management and the hypotensive efficacy of the device during follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Diagnosis of primary or secondary open-angle glaucoma according to the diagnostic criteria of 4th edition of the European Glaucoma Society Guidelines.
3. Need for XEN63 implantation for IOP not controlled by medical therapy, progression of disease or intolerance to topical therapy, in association or not with cataract surgery.
4. Informed consent freely given and obtained before the start of the study.
5. The participant has the ability to understand and the willingness to follow the study instructions and is likely to complete all required visits and procedures.

Exclusion Criteria:

1. Closed-angle glaucoma
2. Previous trabeculectomy or valve or tube placement.
3. Presence of conjunctival scarring, previous conjunctival surgery or other conjunctival pathologies (e.g. pterygium) in the target quadrant.
4. Signs of active inflammation (e.g. blepharitis, conjunctivitis, keratitis, uveitis)
5. Active iris neovascularization or presence of iris new vessels within 6 months of the date of surgery
6. Anterior chamber lenses
7. Presence of intraocular silicone oil
8. Vitreous in anterior chamber
9. Altered episcleral venous drainage (e.g. Sturge Webwer syndrome, nanophthalmos)
10. Known or suspected allergy or sensitization to medications required for the surgical procedure or some component of the device (e.g. glutaraldehyde or porcine derivatives)
11. History of predisposition to the formation of keloids.
12. Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glaucoma patients attending the hospital
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
IOP | up to 2 years
  IOP values before and after 24 months of XEN63 implant.
Number of hypotensive eye drops | up to 2 years
  Number of hypotensive eye drops

SECONDARY OUTCOMES:
IOP | From enrollment to 12 months after surgery
  IOP values before and after 12 months of XEN63 implant.
Number of hypotensive eye drops | From enrollment to 12 months after surgery
  Number of hypotensive eye drops before and after 12 months of XEN63 implant
Complications | up to 2 years
  - Type and number of intraoperative and postoperative complications.
Quality of life after XEN63 implant | up to 2 years
  Quality of life questionnaire (National Eye Institute Visual Function Questionnaire-25) scores over time. The minimum value is 0, the maximum value is 100. Higher score means a better outcome.
Surgical tecnique | during the intervention/procedure/surgery
  Data on surgical technique: site of XEN63 implant
Post operative management | up to 2 years
  Post operative treatment: type of steroids used
Post operative needling | up to 2 years
  Number of needling
Surgical revision | up to 2 years
  Number of surgical revision
Glaucoma Symptom Scale | up to 2 years
  A brief symptom survey specific for persons with glaucoma. This score is transformed to a 0 to 100 scale, with 0 representing presence of a very bothersome problem and 100 representing absence of a problem.
Surgical technique | during the intervention/procedure/surgery
  Data on surgical technique: type of viscoelastic used
Post operative management | up to 2 years
  Type and number of hypotensive drops used to control IOP after surgery if needed.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Oddone, MD, PhD, Principal Investigator — IRCCS-Fondazione GB Bietti
Locations (19):
- Italy (19):
  - Ente ecclesiastico Ospedale Generale Regionale F. Miulli-Acquaviva delle Fonti Bari, Acquaviva delle Fonti, Italy
  - Ospedale della Murgia "Fabio Perinei", Altamura, Italy
  - Ospedale Santa Croce e Carle di Cuneo, Cuneo, Italy
  - SOD Oculistica - AOU Careggi, Firenze, Florence, Italy
  - AUSL di Piacenza UOC Oculistica, Ospedale "Guglielmo da Saliceto, Piacenza, Italy
  - Azienda Ospedaliera Universitaria di Sassari, Dipartimento di Medicina, Chirurgia e Farmacologia Università di Sassari, Sassari, Italy
  - UOC Oculistica Aulss 4, Ospedale di San Donà Di Piave., Venezia, Italy
  - Ospedale S. Andrea, S.O.C. Oculistica, Vercelli, Italy
  - ASST Papa Giovanni XXIII, Bergamo
  - Clinica Oculistica, Ospedale San Giovanni di Dio, Azienda Ospedaliero-Universitaria di Cagliari, Cagliari
  - Clinica Oculistica c/o Azienda Ospedale - Università di Padova, Padua
  - Dipartimento di Scienze Clinico-Chirurgiche, Diagnostiche e Pediatriche, Fondazione IRCCS policlinico San Matteo di Pavia, Pavia
  - Dipartimento di Medicina e Scienze dell'Invecchiamento, Università G.D'Annunzio di Chieti-Pescara, Pescara
  - Clinica Oculistica Universitaria Ospedale Santa Chiara, AOUP-Ospedale Cisanello, Pisa
  - IRCCS-Fondazione GB Bietti, Rome
  - CET Interaziendale AOU Città della Salute e della Scienza di Torino, Torino
  - Ospedale Ca'Foncello AULSS 2 Marca Trevigiana, Treviso
  - Azienda ospedaliera 'C.Panico' Tricase Lecce, Tricase
  - Day service di Oculistica del PPA "F.Fallacara", Triggiano

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fea AM, Menchini M, Rossi A, Posarelli C, Malinverni L, Figus M. Early Experience with the New XEN63 Implant in Primary Open-Angle Glaucoma Patients: Clinical Outcomes. J Clin Med. 2021 Apr 12;10(8):1628. doi: 10.3390/jcm10081628. PMID 33921311
- [Background] Lavia C, Dallorto L, Maule M, Ceccarelli M, Fea AM. Minimally-invasive glaucoma surgeries (MIGS) for open angle glaucoma: A systematic review and meta-analysis. PLoS One. 2017 Aug 29;12(8):e0183142. doi: 10.1371/journal.pone.0183142. eCollection 2017. PMID 28850575
- [Background] Fannin LA, Schiffman JC, Budenz DL. Risk factors for hypotony maculopathy. Ophthalmology. 2003 Jun;110(6):1185-91. doi: 10.1016/S0161-6420(03)00227-6. PMID 12799246
- [Background] Bashford KP, Shafranov G, Shields MB. Bleb revision for hypotony maculopathy after trabeculectomy. J Glaucoma. 2004 Jun;13(3):256-60. doi: 10.1097/00061198-200406000-00015. PMID 15118473
- [Background] Bitrian E, Song BJ, Caprioli J. Bleb revision for resolution of hypotony maculopathy following primary trabeculectomy. Am J Ophthalmol. 2014 Sep;158(3):597-604.e1. doi: 10.1016/j.ajo.2014.05.021. Epub 2014 May 27. PMID 24874999
- [Background] Oyakhire JO, Moroi SE. Clinical and anatomical reversal of long-term hypotony maculopathy. Am J Ophthalmol. 2004 May;137(5):953-5. doi: 10.1016/j.ajo.2003.11.019. PMID 15126172
- [Background] Costa VP, Arcieri ES. Hypotony maculopathy. Acta Ophthalmol Scand. 2007 Sep;85(6):586-97. doi: 10.1111/j.1600-0420.2007.00910.x. Epub 2007 Jun 2. PMID 17542978
- [Background] Jampel HD, Musch DC, Gillespie BW, Lichter PR, Wright MM, Guire KE; Collaborative Initial Glaucoma Treatment Study Group. Perioperative complications of trabeculectomy in the collaborative initial glaucoma treatment study (CIGTS). Am J Ophthalmol. 2005 Jul;140(1):16-22. doi: 10.1016/j.ajo.2005.02.013. PMID 15939389